CLINICAL TRIAL: NCT03917186
Title: Fast-track in Endovascular Aortic Aneurysm Repair With Desflurane and Sevoflurane: a Randomized Clinical Trial
Brief Title: Desflurane vs. Sevoflurane in Endovascular Aortic Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Begoña Quintana Villamandos (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Begoña Quintana Villamandos, Anesthesiologsit, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DESEVAR
Record Dates: First submitted 2017-09-25; First posted 2019-04-16 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Renal Failure
Keywords: Desflurane, Sevoflurane, Endovascular aortic repair
MeSH Terms: conditions — Renal Insufficiency | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group sevoflurane (Active Comparator): Administration under labelling conditions
  Interventions: Drug: Sevoflurane
- Group desflurane (Experimental): Administration under labelling conditions
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — administration of sevoflurane
  Arms: Group sevoflurane
Drug: Desflurane — administration of Desflurane
  Arms: Group desflurane

SUMMARY:
Randomized Clinical Trial following the evaluation of the impact on renal function in patients undergoing endovascular aortic aneurysm repair with two anesthetics protocols (Desflurane versus Sevoflurane) on the first 24 hours after surgery.

DETAILED DESCRIPTION:
Randomized Clinical Trial to evaluate the impact on renal function in patients undergoing endovascular aortic aneurysm repair with two anesthetics protocols (Desflurane versus Sevoflurane) on the first 24 hours after surgery.

Secondary Endpoint: Among secondary endpoints we will evaluate clinical variables such emergence and recovery characteristics (time to extubation and time to emergence-open eyes and response to verbal command), the need for postoperative mechanical ventilation, the post-anesthesia recovery score and ICU length of stay.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years undergoing elective endovascular aortic repair
* who have signed informed consent

Exclusion Criteria:

* urgent surgery
* with known hypersensitivity to Desflurane or Sevoflurane.
* Renal failure in hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Change in Biochemical parameters | All these parameters will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  NGAL in urine
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  Cystatin C(mg/L) in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  Creatinine(mg/dL) in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  sodium(mMol/L) in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  potassium(mMol/L) in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  Chloride(mMol/L) in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  albumin(g/dL) in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  osmolarity(mOsm/Kg) in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  NGAL in plasma
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  Creatinine(mg/dL) in urine
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  sodium(mMol/L) in urine
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  potassium(mMol/L) in urine
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  Chloride(mMol/L) in urine
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  albumin(g/dL) in urine
Change in Biochemical parameters | will be evaluated at baseline (presurgery), at the end surgery and 24 hours after surgery in both study groups
  osmolarity(mOsm/Kg) in urine

SECONDARY OUTCOMES:
Need for postoperative mechanical ventilation | 24 hours
  hours of mechanical ventilation in ICU
ICU length of stay | up to 24 hours
  hours in ICU
anesthetic recovery | These variable will be recorded immediately after surgery (from anesthetics discontinuation). The postanesthesia recovery score before will be recorded at baseline and after surgery. time frame upto 1 hour(stimated)
  time to extubation(minutes).
anesthetic recovery | These variable will be recorded immediately after surgery (from anesthetics discontinuation). The postanesthesia recovery score before will be recorded after surgery. timeframe up to 1 hour(stimated).
  time to spontaneous eye opening(minutes)
anesthetic recovery | These variable will be recorded immediately after surgery (from anesthetics discontinuation). The postanesthesia recovery score before will be recorded after surgery. timeframe up to 1 hour(stimated).
  time until first response to verbal commands(minutes)
anesthetic recovery | These variable will be recorded immediately after surgery (from anesthetics discontinuation). The postanesthesia recovery score before will be recorded at baseline and after surgery. timeframe 1 hour(stimated)
  The post-anesthesia recovery score ( Modified Aldrete score) (0-1-2 from worse to better)

CONTACTS AND LOCATIONS:
Overall Officials: Begoña Quintana, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital general universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Arnalich-Montiel A, Barrio-Perez IM, Burgos-Santamaria A, Fernandez-Riveira C, Lazaro A, Gonzalez-Nicolas MA, Rio J, Bellon JM, Canal MI, Ligero JM, Quintana-Villamandos B. Influence of the type of volatile anesthetic on the development of acute kidney injury after endovascular repair of aortic aneurysm: a randomized controlled trial (DESEVAR study). Front Pharmacol. 2025 Sep 25;16:1660359. doi: 10.3389/fphar.2025.1660359. eCollection 2025. PMID 41079741